CLINICAL TRIAL: NCT03147144
Title: Ultrasonographic Measurements of Uterine Junctional Zone and Association With In Vitro Fertilization Treatment Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0031-17
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasonographic imaging — Ultrasound pelvic scan

SUMMARY:
The aim of this study is to prospectively examine the relationship of the uterine junctional zone thickness, evaluated by ultrasonography and In Vitro Fertilization (IVF) treatment outcome. The study hypothesis is that the uterine junctional zones of women who did not achieve pregnancy will be thicker than those of the women who do achieve pregnancy

DETAILED DESCRIPTION:
Ultrasounds of women who achieve pregnancy after IVF treatment will be compared to ultrasounds of women who do not achieve pregnancy. Their uterine junctional zone thickness will be compared.

The study hypothesis is that the uterine junctional zones of women who did not achieve pregnancy will be thicker than those of the women who do achieve pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF treatment due to male factor, polycystic ovary syndrome and unexplained infertility

Exclusion Criteria:

* Low ovarian reserve
* Having undergone more than one D&C

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women attending the IVF clinic at Hillel Yaffe Medical Center
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Thickened uterine junctional zone | 2 months
  Observed and measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Livna Shafat Heller, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No